CLINICAL TRIAL: NCT01600625
Title: Effects of Minocycline on Cytokine Levels in Severe Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0830
Record Dates: First submitted 2012-05-13; First posted 2012-05-17 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Meibomian Gland Dysfunction
Keywords: meibomian gland dysfunction; inflammatory tear cytokine; minocycline
MeSH Terms: conditions — Meibomian Gland Dysfunction; cyclopia sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline treatment group (Experimental)
  Interventions: Drug: oral minocycline hydrochloride treatment

INTERVENTIONS:
Drug: oral minocycline hydrochloride treatment — Orally received 50 mg minocycline (Minocin, SK chemical, Seoul, Korea) twice a day for 2 months treatment

SUMMARY:
One of the important factors in obtaining successful outcomes when treating severe meibomian gland dysfunction (MGD) is to control the existing ocular and eyelid inflammation. Thus, in previous studies, topical and systemic antibiotics with anti-inflammatory function, such as topical azithromycin, systemic tetracycline, doxycycline and minocycline, have been used to treat severe MGD. In this study, minocycline which had the fewest side effects was used to evaluate the effect on cytokine levels in severe MGD. At study initiation, all patients completed an Ocular Surface Disease Index (OSDI) questionnaire and had an ocular surface, tear, and meibomian gland evaluation that consisted of fluorescein tear break-up time (TBUT), Schirmer test, corneal and conjunctival fluorescein staining, microscopic examination of lid margins and meibomian glands, and tear cytokine levels. All measurements except tear cytokine levels were conducted in the same manner before treatment, after 1 month, and after 2 months of treatment. Tear cytokine levels were evaluated before treatment and after 2 months of treatment. The aim of this research was to determine the concentration of inflammatory cytokines in the tears of patients with MGD and to compare the cytokine levels, corresponding clinical responses, and ocular symptoms before and after 2 months of treatment with oral minocycline.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage 3 or 4 meibomian gland dysfunction
* moderate or marked symptoms of ocular discomfort, itching, or photophobia with limitations of activities
* moderate or severe meibomian gland dysfunction clinical signs
* mild to moderate conjunctival and peripheral corneal staining or increased conjunctival and corneal staining, including central staining
* increased signs of inflammation : moderate or severe conjunctival hyperemia, phlyctenulae

Exclusion Criteria:

* history of previous ocular or intraocular surgery
* evidence of acute or chronic infections or inflammation of the cornea and conjunctiva
* ocular allergy
* autoimmune disease
* history of intolerance or hypersensitivity to any component of the study medications
* use of topical ocular medications
* wearing contact lenses during the study period
* presence of current punctal occlusion
* pregnancy
* lactating women
* children

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
change of inflammatory tear cytokine levels | before treatment and after 2 months of treatment
  Thirty microliters of phosphate-buffered saline will be injected into the inferior conjunctival sac using a micropipette. Approximately 20 μL tear fluid and buffer will be collected with a micropipette.
  Cytokines are measured using the BDTM Cytometric Bead Array (CBA) (BD Bioscience, San Jose, CA). The cytokines analyzed were interleukin (IL)-1β, IL-6, IL-7, IL-8, IL-12p70, IL-17α, interferon-γ (IFN-γ), tumor necrosis factor-α (TNF-α), and monocyte chemotactic protein-1 (MCP-1). Flow cytometry will be performed using the BDTM LSRII system (BD Bioscience, San Jose, CA).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Hom MM, Martinson JR, Knapp LL, Paugh JR. Prevalence of Meibomian gland dysfunction. Optom Vis Sci. 1990 Sep;67(9):710-2. doi: 10.1097/00006324-199009000-00010. PMID 2234831
- [Result] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Result] Knop E, Knop N, Millar T, Obata H, Sullivan DA. The international workshop on meibomian gland dysfunction: report of the subcommittee on anatomy, physiology, and pathophysiology of the meibomian gland. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1938-78. doi: 10.1167/iovs.10-6997c. Print 2011 Mar. No abstract available. PMID 21450915
- [Result] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Derived] Lee H, Min K, Kim EK, Kim TI. Minocycline controls clinical outcomes and inflammatory cytokines in moderate and severe meibomian gland dysfunction. Am J Ophthalmol. 2012 Dec;154(6):949-957.e1. doi: 10.1016/j.ajo.2012.06.009. Epub 2012 Sep 8. PMID 22967863